CLINICAL TRIAL: NCT01975506
Title: An Examination of Occupational Therapy in the Context of Head Start
Brief Title: Occupational Therapy in the Context of Head Start
Status: Completed | Type: Observational
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Other Study IDs: 16898
Record Dates: First submitted 2013-07-29; First posted 2013-11-04 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Developmental Delay
Keywords: Head Start; Occupational Therapy
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- head start practitioners

SUMMARY:
The purpose of this study is to identify the role of occupational therapy within Head Start programs. Representatives within Head Start will be asked to participate in a nationwide internet based survey identifying the amount and type of services provided within this area. The Model of Human Occupation (MOHO) will also be included in the study by identifying current use of the model and how it can be utilized in the future. In order to complete this study to the fullest extent, we must begin by defining the Model of Human Occupation as well as understanding the mission of the National Head Start Association. The vision of MOHO is to support practice that is focused on occupation, client centered, holistic, evidence-based, and complementary to other occupational therapy models. The mission of the National Head Start Association is to coalesce, inspire and support the Head Start field as a leader in early childhood development and education. This has lead researchers to perform the following study: An examination of occupational therapy in the context of Head Start.

DETAILED DESCRIPTION:
Participants will be informed of the intent of the study in the initial e-mail introduction and invitation of participation. Participants will be given the opportunity to ask questions about the study by asking the research assistants, whose names and email addresses will be given. Within the initial email introduction/invitation of participation, participants will be given the name and contact information of the research assistants and will be instructed to direct all questions regarding the survey to them. All data received from the survey participants will be returned de-identified. None of the data collected will be traceable to the survey participants. Participants will be provided the research assistants' email addresses and can contact them should they be interested in receiving any results from the study. The benefits of the study are to advance the overall role of Occupational Therapy services within head start facilities. This study could further understandings of how and / or why certain concepts should / shouldn't be used, could assist administrators in developing quality programming, and contribute to the body of knowledge in Occupational Therapy in Head Start programs. The research assistants' e-mail addresses will be provided in the consent forms with a statement saying that they will be able to contact her via e-mail should they be interested in receiving any results from the study.Informed consent will be obtained through the initial email introduction and formal request for participation. Participants will be provided study information on the first page of the survey and will indicate their consent by clicking "yes" or "no" before beginning the survey.

ELIGIBILITY:
Inclusion Criteria:

Head Start program does not discriminate against gender, so every individual over the age of 18 who works within Head Start programs will be included in this study.

Exclusion Criteria:

Although participants will not be excluded from the study based on ethnicity, non-English speaking individuals will be excluded from this study. Study materials will be presented in English only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals within Head Start programs nationwide will be contacted to participate in an online survey about the use/role of occupational therapy in Head Start. Particapants will be recruited to participate in the study based upon their association with Head Start organizations across the United States. An initial e-mail will be sent to each individual informing them of the purpose of the study, and inviting them to participate in the survey. A link to the survey along with specific instructions in how to complete it will be included in the email. See attached email recruitment script. The age range is from 18 and up because a variety of disciplines may be selected to respond to the survey. Participants under the age of 18 are typically still in school and therefore may lack the exposure and understanding of occupational therapy services and the role of the occupational therapist within the Head Start program.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The Model of Human Occupation(MOHO)Web Based survey | The time commitment for participants will be approximately 15-20 minutes or however long it takes them to complete the online survey
  E-mail will be the primary means of completing this study. Invitation for participation, survey instructions, and survey will all be completed through e-mail.The study will be conducted via the internet through a web based survey program.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bowyer, EdD,MS,OTR, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States